CLINICAL TRIAL: NCT04730492
Title: A Retrospective Observational Study of Hernias Reparation in Patients Who Have Received a Kidney Transplant
Brief Title: HErnias REparation After Kidney Transplantation Study
Acronym: HEREKT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0594
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Prosthesis User; Renal Transplantation
Keywords: renal transplantation; post incision hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Renal Transplantation: Renal Transplantation
- Hernias reparation post renal transplantation: Hernias reparation post renal transplantation

SUMMARY:
Correlation between hernias reparation in patients who have received a kidney transplant. The investigators will analyze the data of patients who have been treated for reparation of incisional hernia after kidney transplantation with or without the placement of a prosthesis.

DETAILED DESCRIPTION:
In the scientific literature, the percentage of post incisional hernia in kidney transplanted patients is very variable, and not too well-argued, especially in the context of prevention and individuation of risk factors.

The increase of surgical management of hernias reparation in renal transplant patients justifies the start of a mon-centric type study. The investigators will look for risk factors with a retrospective, observational study, by analyzing the type of surgical repair of their post-surgical wall defect.

The analysis of costs/benefits on postoperative, intraoperative, or preoperative prevention will be taken into account.

ELIGIBILITY:
Inclusion criteria:

- hernia post renal transplantation

Exclusion criteria:

- underage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have received renal transplantation with post-incisionale hernia
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
disembowelment number in FIG / D | 1 day
  disembowelment number in FIG / D

SECONDARY OUTCOMES:
type of wall closure technique in the context of a kidney transplant | 1 day
  type of wall closure technique in the context of a kidney transplant

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio PANARO, PhD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC